CLINICAL TRIAL: NCT02352727
Title: The Measurement of Nocturnal Hypokinesia in Parkinson's Disease (PD) Patient Compared With Spouse by Wearable Sensors
Acronym: PD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Jirada Sringean, Dr, Chulalongkorn University
Other Study IDs: 153/57
Record Dates: First submitted 2015-01-23; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Parkinson Disease
Keywords: Nocturnal hypokinesia; Accelerometers
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

SUMMARY:
To quantitative measurement of nocturnal hypokinesia of Parkinson's disease patients compares with their spouses by using multisite accelerometers for 1 night at their home. To determine whether the nocturnal movement of Parkinson's disease patients less than normal elderly people or not.

DETAILED DESCRIPTION:
To quantify the severity of nocturnal akinesia, the nocturnal akinesia dystonia and cramp score (NADCS) and Unified Parkinson's Disease Rating Scale (UPDRS) were recorded in the patient group and also details of demographic data, history and physical examinations were included. The patients and spouses wore the 3-axis (x,y,z) accelerometers at bilateral wrists, bilateral ankles, and trunk for 1 night at their home. The 5-minute periods after going to bed and before waking up in the morning were excluded from the analysis. The definition of movement of the trunk is a change of 15 degrees from the previous position and sustained for 5 minutes in any axis. The movement of limbs is defined as a change of 15 degrees from the previous position and sustained for 2 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease patients who met the criteria diagnosis of United Kingdom Parkinson's Disease Society Brain Bank (UKPDSBB) with their spouses which age difference less than 10 years.

Exclusion Criteria:

* 1) patients and/or spouses who were bed ridden,
* 2) a history of other neurological diseases or other muscle and joint diseases,
* 3) no history of hypnotic drug use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: we study the Parkinson's disease patients and their spouses who received the treatment at King Chulalongkorn Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
the number of axial movement of Parkinson's disease patients compare to their spouses defined by accelerometer | one year
the velocity of axial movement of Parkinson's disease patients compare to their spouses defined by accelerometer | one year
the acceleration of axial movement of Parkinson's disease patients compare to their spouses by accelerometer | one year

SECONDARY OUTCOMES:
The correlations between nocturnal hypokinesia parameter (number of axial movement) and severity of Parkinson's disease. | one year
  The correlation between number of axial movement and UPDRS.
The correlations between nocturnal hypokinesia parameter (velocity of axial movement) and severity of Parkinson's disease. | one year
  The correlation between velocity of axial movement and UPDRS.
The correlations between nocturnal hypokinesia parameter (degree of axial movement) and severity of Parkinson's disease. | one year
  The correlation between degree of axial movement and UPDRS.

OTHER OUTCOMES:
The number of nocturia of Parkinson's disease patient | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Stack EL, Ashburn AM. Impaired bed mobility and disordered sleep in Parkinson's disease. Mov Disord. 2006 Sep;21(9):1340-2. doi: 10.1002/mds.20944. PMID 16773640
- [Background] Chaudhuri KR, Schapira AH. Non-motor symptoms of Parkinson's disease: dopaminergic pathophysiology and treatment. Lancet Neurol. 2009 May;8(5):464-74. doi: 10.1016/S1474-4422(09)70068-7. PMID 19375664
- [Background] Verbaan D, van Rooden SM, Visser M, Marinus J, van Hilten JJ. Nighttime sleep problems and daytime sleepiness in Parkinson's disease. Mov Disord. 2008 Jan;23(1):35-41. doi: 10.1002/mds.21727. PMID 17960797
- [Background] Steiger MJ, Thompson PD, Marsden CD. Disordered axial movement in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1996 Dec;61(6):645-8. doi: 10.1136/jnnp.61.6.645. PMID 8971118
- [Background] Bhidayasiri R, Mekawichai P, Jitkritsadakul O, Panyakaew P, Kaewwilai L, Boonrod N, Petchrutchatachart S, Jagota P, Boonpeng K, Singmaneesakulchai S, Setthawatcharawanich S. Nocturnal journey of body and mind in Parkinson's disease: the manifestations, risk factors and their relationship to daytime symptoms. Evidence from the NIGHT-PD study. J Neural Transm (Vienna). 2014 Aug;121 Suppl 1:S59-68. doi: 10.1007/s00702-014-1199-x. Epub 2014 Mar 31. PMID 24682359
- [Background] Salarian A, Russmann H, Vingerhoets FJ, Burkhard PR, Aminian K. Ambulatory monitoring of physical activities in patients with Parkinson's disease. IEEE Trans Biomed Eng. 2007 Dec;54(12):2296-9. doi: 10.1109/tbme.2007.896591. PMID 18075046
- [Background] Yang CC, Hsu YL. A review of accelerometry-based wearable motion detectors for physical activity monitoring. Sensors (Basel). 2010;10(8):7772-88. doi: 10.3390/s100807772. Epub 2010 Aug 20. PMID 22163626
- [Background] Maetzler W, Domingos J, Srulijes K, Ferreira JJ, Bloem BR. Quantitative wearable sensors for objective assessment of Parkinson's disease. Mov Disord. 2013 Oct;28(12):1628-37. doi: 10.1002/mds.25628. Epub 2013 Sep 12. PMID 24030855
- [Result] Weller C, Nicholson PW, Dobbs SM, Bowes SG, Purkiss A, Dobbs RJ. Reduced axial rotation in the spouses of sufferers from clinical idiopathic parkinsonism. Age Ageing. 1992 May;21(3):189-94. doi: 10.1093/ageing/21.3.189. PMID 1615781
- [Result] Weller C, Bowes SG, Kirk CA, Nicholson PW, Dobbs RJ, Dobbs SM. Measurement of axial rotation: its relevance to screening for night-time hypokinesia in old age and parkinsonism. Age Ageing. 1991 Jan;20(1):3-7. doi: 10.1093/ageing/20.1.3. PMID 2028848
- [Result] Godfrey A, Conway R, Meagher D, OLaighin G. Direct measurement of human movement by accelerometry. Med Eng Phys. 2008 Dec;30(10):1364-86. doi: 10.1016/j.medengphy.2008.09.005. Epub 2008 Nov 8. PMID 18996729